CLINICAL TRIAL: NCT03031223
Title: Evaluation of Sensory-motor Response to Low-level Laser Therapy for the Treatment of Spinal Injuries - Protocol for a Randomized, Controlled, Clinical Trial
Brief Title: Evaluation of Sensory-motor Response to Low-level Laser Therapy for the Treatment of Spinal Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Fernanda Cordeiro da Silva, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uni9
Record Dates: First submitted 2016-10-05; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injuries; low-level laser therapy
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-level laser therapy (Experimental): The treatment group will receive LLLT following the protocol outlined below:
  LLLT protocol - radiance will be administered to the injury site transcutaneously at a wavelength of 808 nm using a Twin Flex Evolution diode laser (MMO Equipamento Opto-Eletronicos, Brazil). Twelve sessions will be held (three per week over four weeks). The dose administered to the surface of the skin will be 983 J/cm2 per session, with a treatment area of 4.72 W/cm² and total radiant energy of 25 J. According to the literature, this dose is capable of enhancing functional recovery following an injury.
  Interventions: Radiation: low-level laser therapy
- placebo (Placebo Comparator): laser therapy is applied at low intensity without emitting radiation.
  Interventions: Radiation: low-level laser therapy

INTERVENTIONS:
Radiation: low-level laser therapy — low-level laser therapy

SUMMARY:
Spinal cord injuries have become increasingly frequent due mainly to the increase in urban violence. The growing number of automobile collisions and violence-related events merits particular attention, as such occurrences can lead to death or disability stemming from a spinal injury. The severity of the consequences depends on the location affected and degree of destruction of afferent and efferent spinal cord pathways, with higher, more extensive injuries leading to less physical fitness and functional independence. Unfortunately, injured neurons of the central nervous system are unable to regenerate following a spinal injury and spinal cord regeneration is therefore a major challenge to researchers in the fields of neuroscience and neurologia. Upon receiving an external stimulus, the central nervous system is believed to adapt and reorganize itself using mechanisms to compensate for neuronal loss and promote, even if partially, the remodeling of remaining synaptic connections, leading to new neuronal sprouting. Low-level laser therapy (LLLT) has proven to be a possible option for the stimulation of the repair process in the central nervous system. It is plausible that this type of therapy can offer the same benefits previously established in other types of tissues, the stimulation of bone formation, neovascularization and the regeneration of peripheral nerves. Research groups have investigated the efficacy of LLLT for the treatment of spinal cord injuries and have demonstrated that laser therapy administered simultaneously to an injured sciatic nerve and corresponding segment of the spinal cord accelerates the regeneration process of the injured peripheral nerve.

DETAILED DESCRIPTION:
General objective - Evaluate the effect of LLLT on the sensory-motor response in individuals having suffered a spinal cord injury.

Specific objectives - Investigate the maintenance of the possible sensory-motor response through electromyographic analyses conducted before LLLT and as well as one, 15, 30, 45 and 60 days after the intervention; evaluate functional independence and quality of life in individuals having suffered a spinal cord injury.

Trial design - A randomized, controlled, clinical trial is proposed. displays the flowchart of the development of the study. The trial will be conducted in compliance with the norms governing research involving human subjects and will be submitted for the approval of the Institutional Review Board of University Nove de Julho, São Paulo, Brazil. All participants or their legal guardians will receive clarifications regarding the objectives and procedures of the study and those agreeing to participate will sign a statement of informed consent.

Methods: Participants, interventions and outcomes

Study setting - Physical Therapy Clinics of University Nove de Julho, São Paulo, Brazil Exclusion criteria: complete spinal cord injury, cognitive impairment.

Interventions - The volunteers will be randomly allocated to a control group or treatment group. Evaluations will be conducted before and after the intervention using electromyography of the myotome corresponding to the injured spinal nerve root. The treatment group will receive LLLT following the protocol outlined below:

LLLT protocol - Based on Byrnes et al. and Holanda et al., radiance will be administered to the injury site transcutaneously at a wavelength of 808 nm using a Twin Flex Evolution diode laser (MMO Equipamento Opto-Eletronicos, Brazil). Twelve sessions will be held (three per week over four weeks). The dose administered to the surface of the skin will be 983 J/cm2 per session, with a treatment area of 4.72 W/cm² and total radiant energy of 25 J.

According to the literature, this dose is capable of enhancing functional recovery following an injury.

Recruitment Individuals will be recruited from the physical therapy clinics of University Nove de Julho (São Paulo, Brazil) as well as spinal injury associations, if necessary.

Methods: Assignment of interventions (for controlled trials)

Sequence generation The individuals will be allocated to the different groups based on numbers randomly generated by a computer program.

Allocation concealment mechanism Allocation will be concealed with the use of sealed opaque envelopes. Each envelope will be numbered on the outside and will contain the name of a participant on the inside. The envelopes will be randomly selected using a computer program, with the formation of the control group first, followed by the treatment group.

Implementation The volunteers will be enrolled in the research project of MSc. Fernanda Cordeiro da Silva and the envelopes will be prepared by researcher Paulo Roberto da Costa Palácio. Dr. Sandra Kalil Bussadori will head the project and will run the computer program for the random allocation of the volunteers to the different groups.

Blinding - There will be no blinding.

Methods: Data collection, management and analysis The data will be tabulated and treated using the SPSS 20.0 program for WindowsTM. The data will be submitted to descriptive statistical analysis. The chi-square test and Fisher's exact test will be used to establish the associations of the categorical variables. The Student's t-test will be used for the comparison of mean electromyographic signals. Pearson's correlation coefficients will be calculated for the analysis of the correlation of the continuous variables. The level of significance will be 95% (p < 0.05).

Ethics and dissemination

Research ethics approval - The trial will be conducted in compliance with the norms governing research involving human subjects and will be submitted for the approval of the Institutional Review Board of University Nove de Julho, São Paulo, Brazil. All participants or their legal guardians will receive clarifications regarding the objectives and procedures of the study and those agreeing to participate will sign a statement of informed consent.

Consent or assent - Researchers MSc. Fernanda Cordeiro da Silva and Paulo Roberto da Costa Palácio will present and explain the statement of informed consent to each volunteer. All participants will be informed with regard to the voluntary nature of participation and the possibility of withdrawing from the study at any time with no negative consequences.

Confidentiality - All data collected from the volunteers during the evaluations and treatments will be stored a hard drive to ensure confidentiality.

Declaration of interests - The authors declare no conflicts of interest. Access to data - Only the researchers directly involved in the study will have access to the data.

Ancillary and post-trial care - At the end of the study, all volunteers allocated to the control group will receive LLLT with the same protocol administered to the treatment group to avoid any inequality regarding treatment among the individuals.

Dissemination policy - The findings will be published in scientific journals and presented at conferences on the application of laser therapy and treatment for individuals with spinal injuries.

ELIGIBILITY:
Inclusion Criteria:

* partial spinal injury;
* patients with tetraplegia or paraplegia;
* injury between C3 and L5;
* up to one year elapsed since injury.

Exclusion Criteria:

* complete spinal cord injury;
* cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Electromyography | 15 days after the intervention
  Pre and post-laser electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda C. da Silva, master, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo/SP, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] da Silva FC, Silva T, Gomes AO, da Costa Palacio PR, Andreo L, Goncalves MLL, Fatima Teixeira Silva D, Horliana ACRT, Motta LJ, Mesquita-Ferrari RA, Fernandes KPS, Bussadori SK. Sensory and motor responses after photobiomodulation associated with physiotherapy in patients with incomplete spinal cord injury: clinical, randomized trial. Lasers Med Sci. 2020 Oct;35(8):1751-1758. doi: 10.1007/s10103-020-02968-6. Epub 2020 Apr 26. PMID 32337679
- [Derived] da Silva FC, Gomes AO, da Costa Palacio PR, Politti F, de Fatima Teixeira da Silva D, Mesquita-Ferrari RA, Fernandes KPS, Bussadori SK. Photobiomodulation improves motor response in patients with spinal cord injury submitted to electromyographic evaluation: randomized clinical trial. Lasers Med Sci. 2018 May;33(4):883-890. doi: 10.1007/s10103-018-2447-3. Epub 2018 Feb 13. PMID 29441450